CLINICAL TRIAL: NCT07171957
Title: Investigation of Motor Imagery in Individuals With Chronic Obstructive Pulmonary Disease
Brief Title: Motor Imagery in Chronic Obstructive Pulmonary Disease
Status: Enrolling by invitation | Type: Observational
Sponsor: Kutahya Health Sciences University (Other)
Responsible Party: Principal Investigator, Lütfiye AKKURT, MSc, Principal Investigator, Kutahya Health Sciences University
Other Study IDs: 2025/07-09
Record Dates: First submitted 2025-09-03; First posted 2025-09-15 (Actual); Last update posted 2025-09-15 (Actual); Status verified 2025-09

CONDITIONS: Chronic Obstructive Pulmonary Disease (COPD); Mental Imagery
Keywords: mental imagery; Chronic Obstructive Pulmonary Disease
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- COPD group: Study group
- Control Group: Healthy group

SUMMARY:
The purpose of this study was to compare the motor imagery ability of individuals with Chronic Obstructive Pulmonary Disease (COPD) with those without COPD.

DETAILED DESCRIPTION:
The study will begin after receiving approval from the KSBU Non-Interventional Ethics Committee for its compliance. Before data collection begins, each participant who agrees to the study will be informed about the study, and will be asked to sign a voluntary consent form. After obtaining demographic and disease-specific information, participants will be divided into two groups: COPD and non-COPD individuals, and their cognitive skills, dominant hand preference, and motor imagery abilities will be assessed. The cognitive functions of all participants will be assessed using the Standardized Mini Mental State Examination. Participants will be included in the study if they score ≥24. The dominant hand preference of the participants will be determined using the Edinburgh Hand Preference Questionnaire and recorded on the assessment form. In the tests and surveys to be conducted, the dominant hand will be determined based on the results of this questionnaire, and the results of tests performed with the dominant side will be recorded. The GOLD ABE Assessment Tool will be used to assess COPD patients. As part of the GOLD ABE Assessment Tool, patients' pulmonary function test results, COPD Assessment Test (CAT) results, Modified Health Research Council Dyspnoea Scale (mMRC) results, exacerbation history, and hospitalization history will be recorded. Oxygen saturation values of COPD patients will be recorded. Routine measurement results for oxygen saturation and pulmonary function test values of individuals with COPD will be recorded. Participants' motor imagery skills will be assessed using the Kinesthetic and Visual Motor Imagery Questionnaire-20 (KVIQ-20). The Nine-Hole Peg Test will be used to assess the temporal correspondence between participants' actual and imagined movement (mental chronometry). Temporal correspondence between actual and imagined movement will be calculated using the formula. Participants' mental rotation abilities will be assessed using the hand laterality test (hand identification test), one of the mental rotation subcomponents, using the Recognise Hand mobile application. Data obtained from individuals with COPD and individuals without COPD will be recorded. Based on the data obtained, the motor imagery abilities of the two groups will be compared using appropriate statistical methods. The correlation between the disease-specific knowledge of individuals in the COPD group and their motor imagery abilities will be calculated.

ELIGIBILITY:
Inclusion Criteria:

* Being between 40-70 years of age
* Being diagnosed with COPD
* Having 24 points or more on the Mini Mental State Examination
* Not having a history of acute exacerbation and/or hospitalization in the last month and being clinically stable

Exclusion Criteria:

* Being between 40-70 years old
* Having a score of 24 or above on the Mini Mental State Examination
* Not having any pulmonary, cardiac, orthopedic or neurological disease

Ages: 40 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Chest diseases clinic
Sampling Method: Probability Sample
Enrollment: 188 (Estimated)
Dates: Start 2025-08-01 (Actual); Primary Completion 2026-09-30 (Estimated); Study Completion 2026-12-30 (Estimated)

PRIMARY OUTCOMES:
Kinesthetic and Visual Motor Imagery Questionnaire-20 (KVIQ-20) | Baseline (First assessment)
  Developed to assess imagery ability, the questionnaire aims to determine the extent to which individuals visualize and feel the movements they imagine. The KVIQ-20 consists of 10 visual and 10 kinesthetic items that assess head, shoulders, trunk, upper extremity, and lower extremity movements. All 10 movements are performed in a sitting position. The KVIQ uses a 5-point scale to rate the clarity of imagery (Visual subscale) and the intensity of sensations (Kinesthetic subscale); a score of 5 corresponds to the highest level of imagery and a score of 1 corresponds to the lowest level of imagery. During the test, bilateral assessments are performed. A validity and reliability study for the Turkish version was conducted by Dilek and colleagues. Individuals will be instructed to use a first-person perspective during the MI.

SECONDARY OUTCOMES:
Mental Chronometry Test | Baseline (First assessment)
  The Nine-Hole Peg Test (NHPT) will be used to assess the temporal correspondence between real and imagined movement. The test material consists of nine standard-sized small pegs and a wooden board with nine holes to insert them. The NHPT will be administered with the patient in a sitting position. The patient will be asked to place nine pegs in a box on a table as quickly as possible into the holes of another box, and once completed, immediately remove them and place them back in the same box. The test will be performed with the dominant hand. The test time will be measured with a stopwatch, starting when the hand touches the pegs and ending when the last peg is placed in the box. Subjects will then be asked to imagine performing the NHPT without performing any movement. The time will be started with the command "start," and the subject will mentally imagine the NHPT without actually performing any movement. Upon completion of the test, the time will be stopped when the word "stop" is
Mental Rotation Test | Baseline (First assessment)
  Mental rotation is one of the visual-spatial abilities and can be simply defined as the rotation of objects in 3D. The hand laterality test (hand identification test), one of the subcomponents of mental rotation, will be assessed using the Recognise Hand mobile app. The app was developed and released by NOI Group™. The Recognise Hand app has been shown to accurately measure left-hand-right discrimination and reaction time as part of a stepwise motor imagery rehabilitation program. The app will use a "Vanilla" mode, displaying 20 images at 5-second intervals. Patients will be instructed to respond as quickly as possible whether the image is the right or left hand.

OTHER OUTCOMES:
Edinburgh Handedness Questionnaire | Baseline (First assessment)
  This is a questionnaire used to determine dominant handedness. Individuals mark on the questionnaire which hand they prefer to use during 10 different activities of daily living (drawing, writing, throwing, using scissors, brushing teeth, using a knife, using a spoon, using a broom, lighting a match, and opening a jar). Once the individual has completed their markings, the values for the right and left hands are calculated separately. The left hand score is subtracted from the right hand score, divided by the sum of the right and left hand scores, and the resulting value is multiplied by 100. The total score ranges from 100 to -100. Subjects scoring above 40 are recorded as right-handed; subjects scoring between 40 and -40 are recorded as both-handed; and subjects scoring below -40 are recorded as left-handed. The validity and reliability of the questionnaire in Turkish was conducted by Uysal et al.

CONTACTS AND LOCATIONS:
Overall Officials: Lütfiye AKKURT, Asst.Prof., Study Director — Kütahya Health Sciences University; İlknur KAYA, Asst.Prof., Study Chair — Kütahya Health Sciences University
Locations (1):
- Kütahya Health Sciences University, Kütahya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No